CLINICAL TRIAL: NCT01189552
Title: Depression Treatment for Urban Low Income Minority Substance Users
Brief Title: Depression Treatment for Low Income Substance Users
Acronym: LET'S ACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Stacey Daughters, PhD, Associate Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01DA026424 (NIH); R01DA026424 (NIH)
Record Dates: First submitted 2010-08-24; First posted 2010-08-26 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Substance Use Disorder
MeSH Terms: conditions — Substance-Related Disorders | interventions — Person-Centered Psychotherapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LETS ACT Behavioral Activation Treatment (Active Comparator): LETS ACT is based on the empirically validated Behavioral Activation Treatment for Depression (BAT-D; Lejuez, Hopko, & Hopko, 2001). LETS ACT is based on the belief that the best way to improve mood, remain sober, and to make long-term life changes is by changing and increasing one's activity level. It has been modified to accommodate the needs of a substance using population currently receiving inpatient substance use treatment. Treatment is provided over a 4-week period and is provided in small group format, with each group consisting of 3-5 patients.
  Interventions: Behavioral: LETS ACT Behavioral Activation Treatment
- Nondirective Therapy (NDT) (Placebo Comparator): In NDT, the therapist will create an accepting, nonjudgmental, empathic environment to continuously direct client attention to primary feelings, and to facilitate accepting of affective experience using supportive statements, reflective listening, and empathic communications. Treatment is provided over a 4-week period and is provided in small group format, with each group consisting of 3-5 patients.
  Interventions: Behavioral: Nondirective Therapy (NDT)

INTERVENTIONS:
Behavioral: LETS ACT Behavioral Activation Treatment — LETS ACT is based on the empirically validated Behavioral Activation Treatment for Depression (BAT-D; Lejuez, Hopko, & Hopko, 2001). Treatment includes eight sessions over a four-week period and is provided in small group format, with each group consisting of 3-5 patients.
  Other Names: LETS ACT; Behavioral Activation
  Arms: LETS ACT Behavioral Activation Treatment
Behavioral: Nondirective Therapy (NDT) — The purpose of Nondirective Therapy (NDT) is to provide group therapy interaction, allowing for the development of a close therapeutic relationship and a safe and accepting environment to facilitate change. NDT will be conducted as outlined by Crits-Cristoph (1997). That is, the therapist will create an accepting, nonjudgmental, empathic environment to continuously direct client attention to primary feelings, and to facilitate accepting of affective experience using supportive statements, reflective listening, and empathic communications. Patients will received NDT in a small group format (3-5 participants) and will meet over the course of 4 weeks.
  Other Names: Supportive Counseling
  Arms: Nondirective Therapy (NDT)

SUMMARY:
The objective of the current study is to evaluate the effects of a brief, behavioral activation treatment (the Life Enhancement Treatment for Substance Use; LET'S ACT) on long term outcomes of substance use, HIV risk behaviors and mechanisms of treatment response (depressive symptoms, environmental reward, behavioral activation).

DETAILED DESCRIPTION:
Approximately 22% of substance users suffer from elevated depressive symptoms, which is associated with higher rates of substance abuse treatment dropout, relapse to substance use, and HIV risk behavior. Few interventions targeting reinforcement principles have been developed to meet the specific needs of treatment seeking substance users. One approach that may be especially appropriate in this regard is behavioral activation (BA), which aims to increase individuals' engagement in pleasant events, thereby increasing contact with positive reinforcement and decreasing the frequency of aversive events. BA has been shown to be efficacious in the treatment of depression, and this uncomplicated and straightforward approach may be especially appropriate for the specific needs of an inner city low income substance abusing sample. Further, BA compliments standard substance abuse treatment in several key practical and theoretical ways as it is more easily adopted by staff in these settings, more time efficient (e.g., fewer and shorter sessions, group format), more easily understood by patients who suffer from cognitive limitations due to low education level and chronic drug use, and can incorporate aspects of sobriety into its treatment components. In an initial Stage 1 development project, a version of BA, the Life Enhancement Treatment for Substance Use (LETS ACT), was developed and specifically tailored for inner-city low income minority substance users with elevated depressive symptoms. Results demonstrated that LETS ACT led to a significantly greater reduction in self-reported depressive symptoms and a significant increase in enjoyment and reward value of activities as compared to the TAU control group (Daughters et al., 2008). While preliminary findings prove promising, many questions remain unanswered and several extensions of this work are necessary, including an assessment of post treatment substance use and HIV risk behavior, a contact-matched control, and a larger sample size to allow for more complex analyses of the mechanisms underlying these outcomes. Thus, the objective of the present proposal is to follow-up on our previous Stage 1 treatment development efforts and small scale randomized control trial (RCT) with a fully-powered Stage 2 RCT comparing LETS ACT to nondirective therapy (NDT) among a sample of 263 low income depressed substance users currently receiving residential substance abuse treatment in inner-city Washington, DC.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 65 years of age
* beginning their last month of residential treatment

Exclusion Criteria:

* limited mental competency [Mini Mental State Examination score < 23]
* psychosis
* the use of psychotropic medication for < 3 months
* the inability to give informed, voluntary, written consent to participate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Substance Use | baseline to a 12-month post treatment follow up period
  Urine Screen and Timeline Followback
Beck Depression Inventory (BDI-II; Beck et al., 1996) | BDI-II will be evaluated from baseline to a 12-month follow up period
  The Beck Depression Inventory is a 21-item self-report measure of depressive symptoms.

SECONDARY OUTCOMES:
Behavioral Activation for Depression Scale (BADS) | baseline to a 12-month post treatment follow up period
  level of activation and avoidance behaviors
Reward Probability Index (RPI) | baseline to a 12-month post treatment follow up period
  contact with environmental reward

CONTACTS AND LOCATIONS:
Overall Officials: Stacey B Daughters, Ph.D., Principal Investigator — University of Maryland, College Park
Locations (2):
- United States (2):
  - Salvation Army Harbor Light Treatment Center, Washington D.C., District of Columbia
  - University of Maryland, College Park, Maryland

REFERENCES:
- [Background] Daughters SB, Braun AR, Sargeant MN, Reynolds EK, Hopko DR, Blanco C, Lejuez CW. Effectiveness of a brief behavioral treatment for inner-city illicit drug users with elevated depressive symptoms: the life enhancement treatment for substance use (LETS Act!). J Clin Psychiatry. 2008 Jan;69(1):122-9. doi: 10.4088/jcp.v69n0116. PMID 18312046
- [Derived] Kane L, Benson K, Stewart ZJ, Daughters SB. The impact of spiritual well-being and social support on substance use treatment outcomes within a sample of predominantly Black/African American adults. J Subst Use Addict Treat. 2024 Mar;158:209238. doi: 10.1016/j.josat.2023.209238. Epub 2023 Dec 5. PMID 38061630
- [Derived] Reese ED, Conway CC, Anand D, Bauer DJ, Daughters SB. Distress tolerance trajectories following substance use treatment. J Consult Clin Psychol. 2019 Jul;87(7):645-656. doi: 10.1037/ccp0000403. Epub 2019 Apr 22. PMID 31008636